CLINICAL TRIAL: NCT05490628
Title: The Effects of Cognitive Rehabilitation on Motor Performance, Balance and Fear of Falling in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rüstem Mustafaoğlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUC-omerfarukakan-001
Record Dates: First submitted 2022-07-06; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Cognition Disorder; Fear Anxiety
MeSH Terms: conditions — Stroke; Cognition Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into intervention and control groups. Both groups will be treated for 6 weeks. Each participant will be treated for a total of thirty hours, one hour a day, five days a week.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Traditional exercises:
  stretching exercises, strengthening exercises, balance exercises, walking exercises and fine motor skill exercises.
  Interventions: Other: Conventional Therapy
- Cognitive Rehabilitation Group (Experimental): Cognitive rehabilitation; memory, executive function, attention, concentration and calculation exercises.
  Interventions: Other: Cognitive Rehabilitation; Other: Conventional Therapy

INTERVENTIONS:
Other: Cognitive Rehabilitation — Language, memory, attention and executive function exercises are performed for the participants' deficient cognitive functions.
  Arms: Cognitive Rehabilitation Group
Other: Conventional Therapy — Strengthening, walking, balance and coordination exercises are performed according to the needs of the participants.

SUMMARY:
One of the most common complications in stroke patients is cognitive impairment. Cognitive impairment affects a large part of the life of stroke patients. However, the relationship between cognitive impairment and fear of falling in stroke patients has not been investigated in any study yet. Various treatment approaches have been developed to improve cognitive function. While some of these approaches focus on improving cognitive function, others aim to reach the maximum functional level with various compensation methods taught to the patient in the current cognitive situation. As a result of cognitive interventions, stroke patients' participation in daily life, adherence to treatment and quality of life increase. The aim of this study is to investigate the effects of cognitive interventions on motor performance, balance and fear of falling. This study will contribute to the literature by investigating these effects of cognitive rehabilitation.

DETAILED DESCRIPTION:
Participants will be randomized into two groups as control and experimental groups. The control group will receive traditional rehabilitation intervention, while the experimental group will receive additional cognitive intervention to traditional rehabilitation. Two groups will be evaluated before and after the study. Participants' motor performance, balance and fear of falling will be determined by evaluation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with stroke
* The duration of the disease is in the range of 1-24 months
* Having a score of 21 or lower on the mini mental state test
* Having received 3 or more according to the Functional Ambulation Scale
* Not having a vision problem that will affect the vision of the materials to be used during the treatment
* Being able to communicate sufficiently to understand the simple orders given

Exclusion Criteria:

* Having been diagnosed with bilateral stroke
* Having a neurological disease other than the diagnosis of stroke
* Development of aphasia after stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | a day before the study start
  Developed to evaluate mild cognitive impairments, Montreal Cognitive Assessment assesses different cognitive abilities including executive functions, visuospatial skills, memory, language, attention concentration, abstract thinking, calculation and orientation. It takes about 10 minutes to administer and the highest total score that can be obtained from the test is 30. Accordingly, scores of 21 and above are considered normal.
Montreal Cognitive Assessment | through study completion, an average of 2 months
  Developed to evaluate mild cognitive impairments, Montreal Cognitive Assessment assesses different cognitive abilities including executive functions, visuospatial skills, memory, language, attention concentration, abstract thinking, calculation and orientation. It takes about 10 minutes to administer and the highest total score that can be obtained from the test is 30. Accordingly, scores of 21 and above are considered normal.
Fugl-Meyer Assessment | a day before the study start
  The Fugl-Meyer Assessment is used to evaluate any loss or abnormality in physiological, anatomical structure or function in motor function.
Fugl-Meyer Assessment | through study completion, an average of 2 months
  The Fugl-Meyer Assessment is used to evaluate any loss or abnormality in physiological, anatomical structure or function in motor function.
Tinetti Balance & Gait Test | a day before the study start
  Tinetti Balance and Gait Scale is used to evaluate patients' balance and gait.
Tinetti Balance & Gait Test | through study completion, an average of 2 months
  Tinetti Balance and Gait Scale is used to evaluate patients' balance and gait.
Falls Efficacy Scale International (FES-I) | a day before the study start
  FES-I is a self-report questionnaire that provides information on the level of anxiety about falls for 16 activities of daily living.
Falls Efficacy Scale International (FES-I) | through study completion, an average of 2 months
  FES-I is a self-report questionnaire that provides information on the level of anxiety about falls for 16 activities of daily living.

SECONDARY OUTCOMES:
The Timed Up & Go (TUG) Test | a day before the study start
  TUG is a practical clinical assessment tool developed to measure the physical mobility and motor performance of elderly individuals. TUG measures the time for the person to stand up from the chair, walk 3 meters, and return to the chair and sit.
The Timed Up & Go (TUG) Test | through study completion, an average of 2 months
  TUG is a practical clinical assessment tool developed to measure the physical mobility and motor performance of elderly individuals. TUG measures the time for the person to stand up from the chair, walk 3 meters, and return to the chair and sit.
10 meter walking test | a day before the study start
  10-meter walking test is a practical clinical assessment tool developed to measure walking capacity and motor performance of elderly individuals. The 10-meter walking test is performed by measuring the time it takes for a person to walk at normal walking speed between two markers that are 10 meters apart.
10 meter walking test | through study completion, an average of 2 months
  10-meter walking test is a practical clinical assessment tool developed to measure walking capacity and motor performance of elderly individuals. The 10-meter walking test is performed by measuring the time it takes for a person to walk at normal walking speed between two markers that are 10 meters apart.

CONTACTS AND LOCATIONS:
Overall Officials: Rüstem Mustafaoğlu, Study Director — IstanbulUniversity-Cerrahpasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffmann T, Bennett S, Koh CL, McKenna KT. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2010 Sep 8;2010(9):CD006430. doi: 10.1002/14651858.CD006430.pub2. PMID 20824849
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Niemeijer M, Svaerke KW, Christensen HK. The Effects of Computer Based Cognitive Rehabilitation in Stroke Patients with Working Memory Impairment: A Systematic Review. J Stroke Cerebrovasc Dis. 2020 Dec;29(12):105265. doi: 10.1016/j.jstrokecerebrovasdis.2020.105265. Epub 2020 Sep 11. PMID 32992171
- [Background] Liu TW, Ng GYF, Chung RCK, Ng SSM. Cognitive behavioural therapy for fear of falling and balance among older people: a systematic review and meta-analysis. Age Ageing. 2018 Jul 1;47(4):520-527. doi: 10.1093/ageing/afy010. PMID 29471428